CLINICAL TRIAL: NCT04035746
Title: The Interplay of Microcirculation and Plasticity After Ischemic Stroke
Brief Title: Microcirculation and Plasticity After Stroke
Acronym: IMPreST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC-Nr. 2019-00750
Record Dates: First submitted 2019-07-15; First posted 2019-07-29 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2019-11

CONDITIONS: Stroke, Ischemic
Keywords: Microcirculation; Plasticity; Cohort studies
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-group study: Assessment of microcirculation, brain plasticity and clinical function
  Interventions: Other: Observation of microcirculation and plasticity of the brain

INTERVENTIONS:
Other: Observation of microcirculation and plasticity of the brain — Assessment of microcirculation, brain plasticity and clinical function

SUMMARY:
Reperfusion is the main goal of early medical interventions after stroke, such as thrombolysis and thrombectomy. Recanalization works only if applied early - the earlier the better, but with a statistical cutoff of 4.5 hours where risk of hemorrhage outweighs the benefit. Recently, this cutoff has been put into perspective using standardized perfusion measurements by magnetic resonance imaging (MRI) or computed tomography (CT). Two trials have shown that revascularization is beneficial up to 24 hours after stroke onset if patient selection is based on perfusion imaging. This suggests interindividual differences in the temporal evolution of an infarction. One explanation for interindividual differences is the variability of the collateral blood supply to the brain, which in turn can maintain different perfusion pressures around the infarct core, also called the penumbra region. Insufficient recruitment of these collateral pathways is an independent negative predictor of poor outcome; the insufficiency may in part be explained by insufficient dilatation of arterioles ("low dilator reserve"). So far, interventions to improve collateral perfusion, e.g., induced hypertension, have not demonstrated effectiveness, likely because our understanding of collateral perfusion, demand-dependent dilatation of arteries (cerebrovascular reserve, CVR) and their effect on microcirculation is insufficient.

Functional recovery after a brain lesion is based on plasticity. Plasticity involves the creation of new synapses, fibers (axons and dendrites) and lasting modification to synaptic strength as well as the formation and migration of new neurons. In the cortex surrounding an infarct, plasticity is facilitated by ischemia via modification of gene expression, i.e. a certain time window after stroke, and is stimulated by activity and training. Tissue microcirculatory status and perfusion surrounding the stroke lesion may play a role in the formation of this plasticity. The investigators will analyze the contributions of pre-existing vascular networks, the impact of stroke-affected vessels, timing and degree of recanalization success, brain excitability, and short-term intra-cortical inhibition to better understand how these factors relate to functional recovery after stroke.

ELIGIBILITY:
Inclusion Criteria:

* ≤72h First-ever clinical ischemic stroke at hospital admission
* Occlusion of M1-segment of the middle cerebral artery, and/ or intracranial internal carotid artery, and perfusion deficits with cortical involvement
* 18 years or above
* Living independent before stroke (mRS ≤3)
* Written informed consent of the patient or the when the patient is not able to participate in the consenting procedure, the written authorization of an independent doctor who is not involved in the research project to safeguard the interests of the patient; in that case, post-hoc written informed consent of the patient is needed, or when the patient remains unable to participate in the informed consent procedure, written informed consent of a next of kind

Exclusion Criteria:

* Major cardiac, psychiatric and/ or neurological diseases
* Early seizures
* Known or suspected non-compliance, drug and/ or alcohol abuse
* Contra-indications for Magnetic Resonance Imaging and Transcranial Magnetic Stimulation, such as a history of seizure, prior electroconvulsive therapy, deep brain stimulators or other metal in the head, skull defect, pacemaker; neuroleptic medication; known allergic reaction to contrast material
* Documented evidence that the patient does not want to participate in any scientific study or, in case of lack of documented evidence, no behavior and/or expression(s) that indicate(s) refusal of the patient to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutively admitted to the hospital
Sampling Method: Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in brain microcirculation | <72 hours; 7, 45 and 90 days after stroke onset
  Change in microcirculation of the brain as measured by magnetic resonance imaging (MRI)
Change in brain plasticity | 7, 45 and 90 days after stroke onset
  Change in plasticity of the brain as measured by transcranial magnetic stimulation (TMS)

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale | <72 hours; 7, 45 and 90 days after stroke onset
  Neurological impairments (scale range 0-42, higher values represent a worse outcome)
Fugl-Meyer Motor Assessment - Upper Extremity Subscale | 7, 45 and 90 days after stroke onset
  Upper limb motor function (scale range 0-66, higher values represent a better outcome)
Fugl-Meyer Motor Assessment - Lower Extremity Subscale | 7, 45 and 90 days after stroke onset
  Lower limb motor function (scale range 0-34, higher values represent a better outcome)
Finger extension 1 | <72 hours; 7, 45 and 90 days after stroke onset
  Ability to extend the fingers (scale range 0-2, higher values represent a better outcome)
Finger extension 2 | <72 hours; 7, 45 and 90 days after stroke onset
  Ability to extend the fingers (scale range 0-10, higher values represent a better outcome)
Finger extension 3 | <72 hours; 7, 45 and 90 days after stroke onset
  Ability to extend the fingers (scale range 0-3, higher values represent a worse outcome)
Trunk Control Test | 7 and 90 days after stroke onset
  Trunk ability (scale range 0-100, higher values represent a better outcome)
Functional Ambulation Categories | <72 hours; 7, 45 and 90 days after stroke onset
  Walking ability (independence) (scale range 0-5, higher values represent a better outcome)
Ten-Meter Walk Test | 7, 45 and 90 days after stroke onset
  Gait speed and cadence (scale range is time in seconds, higher values represent a worse outcome)
Modified Rankin Scale | <72 hours; 7, 45 and 90 days after stroke onset
  Global disability (scale range 0-5, higher values represent a worse outcome)
Mobilization | <72 hours; 7 days
  Amount of mobilization (scale range is time in minutes, higher values represent a better outcome)
Concomitant movement therapy | <72 hours; 7, 45 and 90 days after stroke onset
  Intensity of therapy based on charts (scale range is time in minutes, higher values represent a better outcome)
Related Serious Events | <72 hours; 7, 45 and 90 days after stroke onset
  Serious Events (1. death; 2. life-threatening illness or injury; 3. in-patient or prolonged hospitalization; 4. medical or surgical intervention to prevent life threatening illness; 5. led to fetal distress, death or a congenital abnormality or birth defect)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas R Luft, Prof. MD, Study Chair — University of Zurich, University Hospital Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Albers GW, Marks MP, Kemp S, Christensen S, Tsai JP, Ortega-Gutierrez S, McTaggart RA, Torbey MT, Kim-Tenser M, Leslie-Mazwi T, Sarraj A, Kasner SE, Ansari SA, Yeatts SD, Hamilton S, Mlynash M, Heit JJ, Zaharchuk G, Kim S, Carrozzella J, Palesch YY, Demchuk AM, Bammer R, Lavori PW, Broderick JP, Lansberg MG; DEFUSE 3 Investigators. Thrombectomy for Stroke at 6 to 16 Hours with Selection by Perfusion Imaging. N Engl J Med. 2018 Feb 22;378(8):708-718. doi: 10.1056/NEJMoa1713973. Epub 2018 Jan 24. PMID 29364767
- [Background] Carmichael ST, Kathirvelu B, Schweppe CA, Nie EH. Molecular, cellular and functional events in axonal sprouting after stroke. Exp Neurol. 2017 Jan;287(Pt 3):384-394. doi: 10.1016/j.expneurol.2016.02.007. Epub 2016 Feb 10. PMID 26874223
- [Background] Cortes JC, Goldsmith J, Harran MD, Xu J, Kim N, Schambra HM, Luft AR, Celnik P, Krakauer JW, Kitago T. A Short and Distinct Time Window for Recovery of Arm Motor Control Early After Stroke Revealed With a Global Measure of Trajectory Kinematics. Neurorehabil Neural Repair. 2017 Jun;31(6):552-560. doi: 10.1177/1545968317697034. Epub 2017 Mar 16. PMID 28506149
- [Background] El Amki M, Wegener S. Improving Cerebral Blood Flow after Arterial Recanalization: A Novel Therapeutic Strategy in Stroke. Int J Mol Sci. 2017 Dec 9;18(12):2669. doi: 10.3390/ijms18122669. PMID 29232823
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Ginsberg MD. Expanding the concept of neuroprotection for acute ischemic stroke: The pivotal roles of reperfusion and the collateral circulation. Prog Neurobiol. 2016 Oct-Nov;145-146:46-77. doi: 10.1016/j.pneurobio.2016.09.002. Epub 2016 Sep 13. PMID 27637159
- [Background] Mostany R, Chowdhury TG, Johnston DG, Portonovo SA, Carmichael ST, Portera-Cailliau C. Local hemodynamics dictate long-term dendritic plasticity in peri-infarct cortex. J Neurosci. 2010 Oct 20;30(42):14116-26. doi: 10.1523/JNEUROSCI.3908-10.2010. PMID 20962232
- [Background] Nogueira RG, Jadhav AP, Haussen DC, Bonafe A, Budzik RF, Bhuva P, Yavagal DR, Ribo M, Cognard C, Hanel RA, Sila CA, Hassan AE, Millan M, Levy EI, Mitchell P, Chen M, English JD, Shah QA, Silver FL, Pereira VM, Mehta BP, Baxter BW, Abraham MG, Cardona P, Veznedaroglu E, Hellinger FR, Feng L, Kirmani JF, Lopes DK, Jankowitz BT, Frankel MR, Costalat V, Vora NA, Yoo AJ, Malik AM, Furlan AJ, Rubiera M, Aghaebrahim A, Olivot JM, Tekle WG, Shields R, Graves T, Lewis RJ, Smith WS, Liebeskind DS, Saver JL, Jovin TG; DAWN Trial Investigators. Thrombectomy 6 to 24 Hours after Stroke with a Mismatch between Deficit and Infarct. N Engl J Med. 2018 Jan 4;378(1):11-21. doi: 10.1056/NEJMoa1706442. Epub 2017 Nov 11. PMID 29129157
- [Background] Wahl AS, Omlor W, Rubio JC, Chen JL, Zheng H, Schroter A, Gullo M, Weinmann O, Kobayashi K, Helmchen F, Ommer B, Schwab ME. Neuronal repair. Asynchronous therapy restores motor control by rewiring of the rat corticospinal tract after stroke. Science. 2014 Jun 13;344(6189):1250-5. doi: 10.1126/science.1253050. PMID 24926013
- [Derived] Barbagallo M, Zahn M, Zimmermann J, Klovekorn R, Held J, Nemeth B, Reolon B, Bellomo J, Schwarz A, Veerbeek JM, Van Niftrik CHB, Sebok M, Piccirelli M, Michels L, Luft AR, Kulcsar Z, Regli L, Esposito G, Fierstra J, Thurner P, Schubert T, Wegener S. Reperfusion failure after successful thrombectomy of large vessel occlusion stroke: clinical and imaging evidence. Front Neurol. 2025 Aug 22;16:1639880. doi: 10.3389/fneur.2025.1639880. eCollection 2025. PMID 40917674